CLINICAL TRIAL: NCT05651191
Title: A Early Phase 1 Clinical Trial To Evaluate the Safety and Efficacy of Human CD19 Targeted DASH CAR-T Cells Injection for Subjects With Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia
Brief Title: To Evaluate the Safety and Efficacy of Human CD19 Targeted DASH CAR-T Cells Injection for Subjects With R/R B-ALL
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hrain Biotechnology Co., Ltd. (Industry)
Collaborators: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRAIN01-ALL04-POC
Record Dates: First submitted 2022-12-02; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: CD19; CAR-T; B-cell acute lymphoblastic leukemia; Relapsed /Refractory
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human CD19 Targeted DASH CAR-T Cells Injection (Experimental): Single administration：0.5×10^6 CAR+T, 1.0×10^7 CAR+T, 2.0×10^7 CAR+T
  Interventions: Drug: Human CD19 Targeted DASH CAR-T Cells Injection

INTERVENTIONS:
Drug: Human CD19 Targeted DASH CAR-T Cells Injection — Autologous genetically modified anti-CD19 CAR transduced T cells
  Other Names: CD19 DASH CAR-T

SUMMARY:
This study is a single-arm, open-label, dose-escalation trial to explore the safety, tolerability and pharmacokinetic/pharmacodynamics characteristics of human CD19 targeted DASH CAR-T Cells injection, and to preliminarily observe the efficacy of the trial drug in patients with relapsed/refractory B-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
Subjects with relapsed/refractory B-cell acute lymphoblastic leukemia can participate if all eligibility criteria are met. Tests required to determine eligibility including disease assessments, a physical exam, Electrocardiograph, Computed tomography（CT）/Magnetic Resonance Imaging(MRI)/Positron Emission Tomography（PET）, and blood draws. Subjects will receive preconditioning chemotherapy prior to the infusion of human CD19 targeted DASH CAR-T Cells injection. After the infusion, subjects will be followed for adverse events, pharmacokinetic/pharmacodynamics characteristics, efficacy of human CD19 targeted DASH CAR-T cells. Study procedures may be performed while hospitalized.

ELIGIBILITY:
Inclusion Criteria:Subjects must meet all of the following criteria to be enrolled:

* 18 to 70 years old (including cut-off value), Male and female;
* Expected survival > 12 weeks;
* ECOG score 0-1;
* Bone marrow examination clearly diagnosed as B-cell acute lymphoblastic leukemia, CD19 positive, and who met one of the following conditions:

  1. Those who failed to achieve CR after at least 2 courses of standard chemotherapy or had early relapse after complete remission (<12 months) or late relapse after complete remission (≥ 12 months) and failed to achieve CR after 1 course of standard chemotherapy;
  2. For Ph+ ALL: in addition to receiving at least 2 courses of standard chemotherapy, at least two TKIs should be treated with no complete remission or relapse after complete remission; (Patients who cannot tolerate TKI therapy or have TKI treatment contraindications or have T315i mutation are excluded);
  3. Those who relapse after stem cell transplantation are not affected by previous treatments;
* The venous access required for collection can be established and leukapheresis can be carried according to the judgement of investigators;
* Liver, kidney and cardiopulmonary functions meet the following requirements:

  1. Serum creatinine ≤ 1.5×ULN;
  2. Left ventricular ejection fraction > 50%;
  3. Baseline oxygen saturation > 96%;
  4. Total bilirubin ≤ 2×ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3×ULN (As judged by the investigator, the elevation of transaminase caused by the ALL disease itself, ALT and AST ≤ 5×ULN);
* Able to understand and sign the Informed Consent Document.

Exclusion Criteria:Any one of the following conditions cannot be selected as a subject：

* Graft-versus-host disease (GVHD), or need to use immunosuppressants after transplantation;
* Patients with hyperleukocytosis (white blood cell count ≥ 50×10^9/L) or whose disease progressed rapidly according to the investigator's judgment at the time of enrollment and cannot ensure the completion of a complete treatment cycle;
* Malignant tumors other than acute lymphoblastic leukemia within 5 years prior to screening, in addition to adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical resection, ductal carcinoma in situ after radical resection and thyroid cancer after radical resection;
* Subjects with positive Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) and peripheral blood hepatitis B virus (HBV) DNA titer detection higher than the lower limit of the research center can detect; hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive; human immunodeficiency virus (HIV) antibody positive; syphilis detection positive;
* Any instability of systemic disease, including but not limited to unstable angina, cerebrovascular accident, or transient cerebral ischemic (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York heart association (NYHA) classification ≥ III), need drug therapy of severe arrhythmia, liver, kidney, or metabolic disease;
* Active or uncontrollable infection requiring systemic therapy within 14 days prior to enrollment;
* Pregnant or lactating woman, and female subject who plans to have a pregnancy within 1 year after cell transfusion, or male subject whose partner plans to have a pregnancy within 1 year after cell transfusion;
* Received CAR-T treatment or other gene therapies before enrollment;
* Patients with symptoms of central nervous system;
* Subjects who are receiving systemic steroid treatment and requiring long-term systemic steroid treatment during the treatment as determined by the investigator before screening (except inhalation or topical use);
* The investigators consider other conditions unsuitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity (DLT) | 28 days post infusion
  Safety Indicators

SECONDARY OUTCOMES:
Pharmacokinetics parameters - the highest concentration of Human CD19 Targeted DASH CAR-T Cells amplified in peripheral blood after reinfusion | 2 years post infusion
  Effectiveness Metrics
Pharmacokinetics parameters - the time to reach the highest concentration of Human CD19 Targeted DASH CAR-T Cells amplified in peripheral blood after reinfusion | 2 years post infusion
  Effectiveness Metrics
Pharmacokinetics parameters - the 28-day area under the curve of Human CD19 Targeted DASH CAR-T Cells amplified in peripheral blood after reinfusion | 2 years post infusion
  Effectiveness Metrics
Pharmacodynamics characteristics - the detection values of IL-6, IFN-γ, IL-15 cytokines in peripheral blood | 2 years post infusion
  Effectiveness Metrics
Overall response rate (ORR, include CR and CRi) after administration | 3 months post infusion
  Effectiveness Metrics
Duration of remission (DOR) after administration | 2 years post infusion
  Effectiveness Metrics
Overall Survival (OS) after administration | 2 years post infusion
  Effectiveness Metrics

CONTACTS AND LOCATIONS:
Overall Officials: Qingming Wang, M.D., Principal Investigator — Second Affiliated Hospital of Nanchang University
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No